CLINICAL TRIAL: NCT03890185
Title: Randomized Phase II Trial of Docetaxal and Cisplatin Versus Low-Dose Fractionated Radiation Plus Docetaxal and Cisplatin as Induction Therapy in Locally Advanced Nasopharyngeal Cancer
Brief Title: Docetaxal & Cisplatin vs LDFRT + Docetaxal & Cisplatin in Locally Advanced NPC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2121 063
Record Dates: First submitted 2019-01-16; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-01

CONDITIONS: Nasopharyngeal Cancer
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Drug Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Chemo+RT low dose (Experimental): Chemo + Low dose RT: Intervention will include chemotherapy using Docetaxel 75mg/m2 IV D1, Cisplatin (CDDP) 75mg/m2 IV D1 and radiation therapy (LDFRT) using 50 cGy of radiation per fraction BID on the day of chemotherapy and the day after during induction i.e. 50 cGy x 4 times per cycle given for a total of 2 cycles every 21 days.
  Interventions: Combination Product: Chemo + Low dose RT; Drug: Chemo alone
- B: Chemo alone (Active Comparator): Chemo alone: Intervention will include chemotherapy using Docetaxel 75mg/m2 IV D1 and Cisplatin (CDDP) 75mg/m2 IV D1 given for 2 cycles every 21 days.
  Interventions: Combination Product: Chemo + Low dose RT; Drug: Chemo alone

INTERVENTIONS:
Combination Product: Chemo + Low dose RT — Intervention will include chemotherapy using Docetaxel 75mg/m2 IV D1, Cisplatin 75mg/m2 IV D1.Radiathion therapy (LDFRT) using 50 cGy of radiation per fraction BID on the day of chemotherapy and the day after during induction i.e. 50 cGy x 4 times per cycle given for total of 2 cycles every 21 days.
  Other Names: Chemotherapy, Low Dose Radiation Therapy
Drug: Chemo alone — Chemo alone: Intervention will include chemotherapy using Docetaxel 75mg/m2 IV D1 and Cisplatin (CDDP) 75mg/m2 IV D1 given for 2 cycles every 21 days.
  Other Names: Chemotherapy

SUMMARY:
The central hypothesis is to test Low Dose Fraction Radiotherapy (LDFRT), as a potentiator of Docetaxel and Cisplatin efficacy in locally advanced nasopharyngeal cancer.

DETAILED DESCRIPTION:
Nasopharyngeal cancer is the commonest cancer of the head and neck in Saudi Arabia and constitutes nearly a half (44%) of all head and neck cancers diagnosed annually according to the National Cancer Registry Data. Majority of our patients present with locally advance disease which adversely affect their treatment outcome. The treatment of this disease has evolved over the last several years and several Phase III trials have now shown that combined chemotherapy and radiation are significantly superior to treatment with radiation therapy alone. However, results for treatment of the Stage III and IV disease remains less than satisfactory with a 5-year survival of 60-70 %. Recent data in other head and neck cancer sites including nasopharyngeal cancer indicates that the use of chemotherapy in combination with radiation may improve the outcome of therapy primarily by a reduction in the rate of distant metastasis. Induction chemotherapy alone has, however, failed to show an improvement in survival compared to radiation therapy alone. The administration of induction chemotherapy followed by concurrent chemo-radiation appears the most promising approach. Our experience at KFSH&RC with induction chemotherapy followed by chemo-radiation in Stage IV cancers, still reveals that approximately 25- 30% of patients will develop local relapse in the nasopharyngeal site; and 35- 40 % of patients are likely to develop distant metastasis. The most promising recent schedule of induction chemotherapy has been the use of Docetaxel and Cisplatin followed by concurrent Cisplatin and radiation. A recent Phase II study demonstrated that the three-year progression-free survival and overall survivals was improved with the use of this induction regimen. A variety of treatment strategies are currently being investigated in hope of achieving improved local control and enhanced survival of patients. These include addition of new chemotherapy drugs, other targeted agents such as Bevacizumab, Cetuximab, etc and radiation fractionation. The rationale for using neoadjuvant chemotherapy is that a reduction in the overall tumor burden will permit more effective local therapy and reduce the rates of distant metastases. Neoadjuvant cisplatin / docetaxel are active agents for locally advanced nasopharyngeal cancer. The addition of docetaxel to platinum containing neoadjuvant chemotherapy in other locally advanced head and neck squamous-cell carcinoma have also been shown to improve survival.

ELIGIBILITY:
Inclusion Criteria:

1. WHO II-III carcinoma of the nasopharynx, histologically proven.
2. Locally advanced stage III and IV (minimal intracranial extension only) with absence of distant metastases.
3. Age between 18 and 70 years.
4. ECOG performance status 0-2.
5. Hematological function parameters performed within 10 days before inclusion:

   * Neutrophils ≥ 1000 * 109/l.
   * Platelets: ≥ 100 * 109/l.
   * Hemoglobin: ≥ 9 g/dl
6. Adequate hepatic function, defined as follows within 2 weeks prior to registration:

   * Total bilirubin is normal
   * AST (SGOT) and ALT (SGPT) <= 2.5 * upper limit of normal (ULN) of each center.
   * Alkaline phosphatase <= 2.5 * ULN.
7. Renal function parameters performed within 10 days before inclusion: normal serum creatinine and creatinine clearance must be ≥ 55 ml/min.
8. Patient who has given his/her written consent before any specific procedure of the protocol.

Exclusion Criteria:

1. Patients who present stage I, IIa, IIb and IVc.
2. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease-free for a minimum of 3 years (e.g., carcinoma in situ of the breast, oral cavity, or cervix are all permissible);
3. Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is permitted;
4. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields.
5. Head and neck surgery of the primary tumor or lymph nodes prior to registration, with the exception of incisional or excisional biopsies.
6. Patients receiving other experimental therapeutic cancer treatment;
7. Blood pressure at baseline > 150/100 mmHg;
8. Peripheral neuropathy CTCAE, v. 4.0 h grade 2
9. Severe, active co-morbidity, defined as follows:

   * Major medical or psychiatric illness, which in the investigators' opinion would interfere with the completion of therapy and follow up or with full understanding of the risks and potential complications of the therapy.
   * Unstable angina and/or congestive heart failure or peripheral vascular disease requiring hospitalization within the last 12 months, or other cardiac compromise that in the judgment of the investigator will preclude the safe administration of a study drug.
   * Acquired Immune Deficiency.
   * Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
   * Prior allergic reaction to the study drug(s) involved in this.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of chemo and radiation toxicities | Three years
  Chemotherapy and acute radiation toxicities as evaluated using the revised NCI (CTCAE) Version 4.03

SECONDARY OUTCOMES:
Distant and loco regional failure | Three years
  Distant and loco regional failure as evaluated using Response Evaluation Criteria in Solid Tumors (RECIST)

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Alrajhi, MD, Principal Investigator — King Faisal Specialist Hospital & Research Center

IPD SHARING:
Plan to Share IPD: No